CLINICAL TRIAL: NCT00573118
Title: A Retrospective Analysis of Possible Association Between Severe Pregnancy Complications and Elevated Factor VIII Plasma Activity.
Brief Title: Severe Pregnancy Complications Are Associated With Elevated Factor VIII Plasma Activity
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Eli Rimon,MD, Tel Aviv medical center; Israel
Other Study IDs: FactorVIII
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2007-12

CONDITIONS: Pregnancy Complications; Preeclampsia; Placental Abruption; Intrauterine Fetal Growth Restriction; Intrauterine Fetal Death
Keywords: Pregnancy complications: preeclampsia , severe IUGR , IUFD or placental abruption (n = 5).
MeSH Terms: conditions — Pregnancy Complications; Pre-Eclampsia; Abruptio Placentae; Stillbirth; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: The study group included 49 patients with a previous history of one or more of the following pregnancy complications: preeclampsia (n = 17), severe IUGR (n = 13), IUFD (n = 14) or placental abruption (n = 5).
- 2: The control group included 49 healthy women who delivered during the study period, who did not smoke during pregnancy and in whom pregnancy and delivery were uneventful

SUMMARY:
Congenital and acquired thrombophilia were identified as risk factors for thrombosis in systemic vessels.Thrombophilias have also been recently found to be associated with preeclampsia, intrauterine fetal growth restriction (IUGR), placental abruption, intrauterine fetal death (IUFD) and repeated pregnancy loss.These severe pregnancy complications are thought to result from thrombotic events occurring in the uteroplacental circulation. Accumulating data have established an association between elevated plasma activity of factor VIII and thrombosis although the mechanism is still not defined and elevated factor VIII activity is now regarded as being equivalent to thrombophilia.

We intend to investigatthe association between factor VIII levels and severe pregnancy complications which are considered to result from placental vascular pathology, i.e., preeclampsia, IUGR, placental abruption and IUFD. We hypothezise that the prevalence of elevated factor 8 will be higher among women with pregnancy complications compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* Women who had either normal pregnancy or complicated pregnancy.

Exclusion Criteria:

* Other causes of pregnancy complication such as infections, anomalies and fetal malformations

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women who had either normal pregnancy or complicated pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2000-01; Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
prevalenc of elevated factor VIII | RETROSPECTIVE

CONTACTS AND LOCATIONS:
Overall Officials: Eli Rimon, MD, Principal Investigator — Tel Aviv medical center,Israel
Locations (1):
- Tel Avis sourasky medical center, Tel Aviv, Israel